CLINICAL TRIAL: NCT00430430
Title: Lipoprotein Turnover on Low- and High-MUFA Portfolio Diets
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Toronto (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, David Jenkins, Principle Investigator, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REB 05-120
Record Dates: First submitted 2007-01-30; First posted 2007-02-01 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2016-10

CONDITIONS: Hyperlipidemia; Cardiovascular Diseases; Diet Therapy
MeSH Terms: conditions — Hyperlipidemias; Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- High MUFA (Experimental): high monounsaturated fat background diet to portfolio diet
  Interventions: Procedure: High MUFA dietary portfolio
- Low MUFA (Active Comparator): low monounsaturated fat background diet to portfolio diet
  Interventions: Procedure: Low MUFA dietary portfolio

INTERVENTIONS:
Procedure: High MUFA dietary portfolio — high monounsaturated fat background diet to dietary portfolio
  Arms: High MUFA
Procedure: Low MUFA dietary portfolio — low monounsaturated fat background diet to dietary portfolio
  Arms: Low MUFA

SUMMARY:
Low and very low carbohydrate diets, such as the Atkins' Diet, have recently gained attention for their potential health benefits from weight loss and have gained some scientific support from a growing number of studies. Benefits have been noted in relation to raised "good" cholesterol, lower "bad" cholesterol and triglycerides. Other studies have shown an advantage in substituting vegetable fat for carbohydrate in insulin resistant individuals and in some instances in type 2 diabetes where improvements were seen in "good" cholesterol and blood sugars. At the same time, our research have been exploring diets containing less processed carbohydrates and other components which in combination (portfolio diet) have a similar cholesterol lowering effect to drug therapy.

Therefore we wish to determine whether our cholesterol-lowering components (portfolio diet) should be incorporated into lower carbohydrate diets especially to preserve "good" cholesterol and lower "bad" cholesterol for decreasing the risk of heart disease.

DETAILED DESCRIPTION:
All subjects will undergo two parallel 2-phase treatments. On one treatment, subjects will be placed on a low fat diet for one month (control run-in diet) and then for the second month will continue on the low- fat diet (i.e. low-MUFA) with the addition of the portfolio components. The order of these two phases will not be randomized. The other treatment will be similar to the above except that the background diet of the portfolio phase will be high in monounsaturated fat (high-MUFA). Subjects will be allocated randomly to either treatment. Diets will be metabolically controlled and all food will be provided at weekly intervals.

Subjects will come after a 12h overnight fast to the Risk Factor Modification Center at St. Michael's Hospital or the Department of Nutritional Sciences, University of Toronto immediately prior to commencement of each treatment phase and at weekly intervals during the course of each study period. Prior to the start of the study, subjects will be instructed on details of the study diet protocol. They will also be asked to maintain a constant level of physical activity throughout the course of the study. At all visits, body weight (in kg) will be obtained in indoor clothing, without shoes, and blood pressure will be taken twice in the dominant arm after subjects have been seated for at least 20 minutes. Height (in cm) will be recorded at the first visit. Throughout the study period, subjects will maintain the diet prescribed on their initial visit. At every other visit of each treatment phase, subjects will provide a fasting blood sample. The kinetic tests of lipoprotein metabolism will be performed during the 4th and 8th week of the study. At baseline and during the last week of each study phase, 24h urine collection and 12h breath hydrogen collections will be completed.

The measurement of apolipoprotein in vivo kinetics will be carried out using a primed-constant infusion of [D3]L-leucine. This protocol allows for the determination of the kinetics of all apolipoproteins simultaneously. Kinetics studies will be conducted in the constantly fed state where participants receive 1/30th of their daily energy requirements every half-hour for the whole duration of the test (15 hours). These methods are described in detail in previous publications from our group. Briefly, at 7am on the morning of the study, after a 12-hour overnight fast, participants will be admitted to the Toronto General Hospital Clinical Investigation Unit and two intravenous catheters (IV's) will be inserted, one into each forearm vein. One IV will be for infusion of the stable isotope described below and one for withdrawal of blood samples. After achieving a steady state (3hrs after the small half-hourly meals), subjects will first receive a bolus injection of 10 µmol/kg of body weight of [D3]L-leucine ([D3]L-leucine 98%, C/D/N Isotopes) dissolved in physiological saline (0.9% NaCl) and then a constant infusion of 10 µmol/kg/h of [D3]L-leucine for 12 hours via an intravenous line inserted into a left forearm vein. Blood samples will be collected at regular intervals (0, 1/2, 1, 2, 4, 6, 8, 10, 11, 12hrs). All lipoprotein subfractions will be separated by sequential ultracentrifugation and frozen thereafter at -80oC until they are processed for analysis.

ELIGIBILITY:
Inclusion Criteria:

* men and postmenopausal women
* Body mass index > 18.5 kg/m2 and < 40 kg/m2
* Fasting plasma triglyceride (TG) concentration > 2.5 mmol/l and < 6.0 mmol/l at recruitment.
* Fasting plasma LDL cholesterol concentration > 3.4 mmol/l at recruitment.
* Fasting plasma HDL cholesterol concentration < 1.0 mmol/l at recruitment.
* living within a 40 km radius of St. Michael's Hospital.

Exclusion Criteria:

* Premenopausal women will be excluded due to the fluctuation of blood lipids during the menstrual cycle and the difficulty of synchronising the timing of three one month studies with the same point in the menstrual cycle.
* Taking cholesterol medications at the start of the study. However, with their physician's approval those who wish to join but are already taking cholesterol-lowering medications (or cholesterol lowering natural health products) may join the study providing the medications (or natural health products) are stopped for at least 2 weeks before starting the study and throughout the study.
* Patients with uncontrolled high blood pressure will be excluded. The cut off for raised blood pressure has been taken as greater than 140/90mmHg. Patients with systolic blood pressure between 140-150mmHg and diastolic blood pressure between 90-95mmHg may be accepted, since we have found that on the diet their blood pressures tend to be lowered into the acceptable range. For patients in the above normal range (as above), a letter will be required from the physician responsible for their care.
* Changing the type or dose of their drug treatment during the study.
* Those judged as having a likelihood of being non-compliant with instructions for whatever reason. Those with low compliance to lipid-lowering therapy will not be selected.
* Food allergies
* Evidence or history of diabetes, renal liver disease or gastrointestinal disease. Patients will be excluded if they have gross xanthoma or advanced premature cardiovascular disease since this group may include hyperabsorbers of plant sterols.
* Patients with major cardiovascular event (stroke or myocardial infarction), with secondary causes of hypercholesterolemia (or untreated hypothyroidism), with uncontrolled blood pressure, major disability or disorder such as liver disease, renal failure or with major surgery < 6 months prior to randomization. Individuals predisposed to hemorrhagic stroke (on the basis of untreated raised blood pressure) will also be excluded.
* Antibiotic use within the last three months.
* Hormone replacement therapy.
* Smokers or have significant alcohol intake (>1 drink/d).
* Disallowed medications will be cholesterol lowering drugs which if prescribed by patients' physicians while on the study will be a reason for discontinuation from the study. Introduction of cholesterol lowering natural health products during the study will also be a reason for withdrawing a participant from the study.
* individuals with acute (<6 weeks) or chronic (>6 weeks) infections, either bacterial or viral, or individuals suffering from chronic inflammatory diseases

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2007-04; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
HDL-C and VLDL-TG, synthesis and fractional catabolic rates of their respective apolipoproteins, apo AI and B100 | 2 months

SECONDARY OUTCOMES:
LDL-C, LDL particle size, total and VLDL triglyceride, C-reactive protein, intravascular enzymes, HDL subfractions, blood glucose and insulin (HOMA models S and B), and relation of listed outcomes to kinetic parameters | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: David JA Jenkins, MD, PhD, DSc, Principal Investigator — University of Toronto and St. Michael's Hospital
Locations (1):
- Risk Factor Modification Centre, St. Michael's Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Jenkins DJ, Chiavaroli L, Wong JM, Kendall C, Lewis GF, Vidgen E, Connelly PW, Leiter LA, Josse RG, Lamarche B. Adding monounsaturated fatty acids to a dietary portfolio of cholesterol-lowering foods in hypercholesterolemia. CMAJ. 2010 Dec 14;182(18):1961-7. doi: 10.1503/cmaj.092128. Epub 2010 Nov 1. PMID 21041432